CLINICAL TRIAL: NCT05983549
Title: The Effect of Neutral Versus Liberal fLuId Balance In TraumaTic Brain Injury: a Randomised Phase II Feasibility Controlled Trial
Brief Title: Neutral Versus Liberal fLuId In Traumatic Brain Injury: a Randomised Controlled Trial
Acronym: LIMIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Chiara Robba, Researcher, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-07-12; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Traumatic Brain Injury; Fluid Overload; Outcome, Fatal
MeSH Terms: conditions — Brain Injuries, Traumatic; Edema | interventions — Water-Electrolyte Balance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be blinded in knowing the arm, outcome assessors will be not involved in the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (No Intervention): Patients will receive fluids according to clinical practice
- Neutral balance (Active Comparator): Patients will receive fluids aiming to a neutral balance
  Interventions: Procedure: fluid balance

INTERVENTIONS:
Procedure: fluid balance — patients will receive fluids with the aim to achieve a neutral balance
  Arms: Neutral balance

SUMMARY:
Feasibility and safety of targeting neutral vs liberal fluid balance in traumatic brain injured patients: a phase II randomized controlled trial

DETAILED DESCRIPTION:
To determine whether a zero fluid balance strategy during the first week compared to a more liberal fluid policy (allowing positive balance) is feasible in adult intensive care unit (ICU) patients with traumatic brain injury (TBI).Participants randomized to neutral fluid balance will be assessed daily with the aim to maintain a mean daily fluid balance of 0 over the course of the first 5 days from randomization (maximum at day 7 of ICU stay). In case of need for augmentation of cerebral perfusion pressure with 0 balance, fluids will be allowed according to a predefined protocol (see further).Participants randomized to the control group will receive the standard fluid management required as determined by the treating team. Fluid strategy as randomised should be applied for at least 5 days from randomization.

Primary aim: ● Feasibility: ability to achieve a daily neutral balance (0 +/- 500 ml) in the intervention group.

Secondary aims:● Incidence of renal complications, including acute kidney injury, need for renal replacement, multiorgan failure

* Respiratory complications including reduced partial pressure of oxygen/ fraction of inspired oxygen (P/F) ratio
* Cardiopulmonary complications, i.e myocardial infarction, cardiac failure, cardiac arrhythmias, ventricular or supraventricular, pulmonary oedema, ventilator associated pneumonia, acute respiratory distress syndrome
* Difference in mean and daily CPP among the groups
* Difference in daily fluid balance and fluid input during the first 7 days after ICU admission
* Total and daily dose of vasopressors and diuretics during ICU stay
* Vasopressor-free days up to 28 days from ICU admission
* ICU-free days up to 28 days
* Ventilator-free days up to 28 days from intubation.
* Maximum Therapy intensity level (TIL) during the 5 days of randomization

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with TBI (isolated or with extracranial injuries, with and without ICP monitoring)
* Admitted to intensive care unit
* Age >18 years
* Enrolment <48h after ICU admission

Exclusion Criteria:

* Enrolled in another clinical trial that is unapproved for co-enrolment
* Pregnant or suspected pregnancy
* Concomitant hemorrhagic shock expected to require surgical treatment in the following 24h from inclusion or requiring polytransfusions (> 6 blood products or massive transfusion protocol)
* Hemodynamic instability (HR > 120 despite fluid resuscitation of at least 1 liter, and systolic blood pressure < 90 mmHg) at the ICU admission requiring high dosage of norepinephrine (> 0.5 mcg/kg/min) or inotropes (any dose)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility- rate of patients able to achieve neutral fluid balance( 0 +/- 500 ml) during the first week from ICU admission | 7 days
  Ability to target and achieve a daily and total neutral fluid balance (0 +/- 500 ml) in the intervention group. In particular,testing the hypothesis of whether all pairwise differences between group means are the same in a design of repeated measures with 7 days points. We hypothesise a mean of 0 ml in the conservative group, a mean of 1000 ml in the liberal group and standard deviation in the population of 850 ml (500 ml in the conservative group and 1000 ml in the liberal group)

SECONDARY OUTCOMES:
Safety to achieve neutral balance, i.e. the estimation of the difference of incidence of renal, pulmonary, cardiac complications between the two arms | From date of randomization until the date of intensive care unit discharge or death assessed up to 6 months
  Complications occurring during the ICU stay
Rates of patients who die and experience poor neurological outcome after 6 months from ICU admission | 6 months from ICU admission and enrolment
  at 6 months, at hospital and ICU discharge

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available
Supporting Information: Study Protocol